CLINICAL TRIAL: NCT01737775
Title: Comparative Ultrasonic Study of Post Operative Diaphragmatic Dysfunction in Abdominal and Head and Neck Surgery
Acronym: Under the Dome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012.718
Record Dates: First submitted 2012-11-23; First posted 2012-11-30 (Estimated); Last update posted 2013-08-09 (Estimated); Status verified 2013-08

CONDITIONS: Diaphragmatic Dysfunction
Keywords: diaphragmatic dysfunction; ultrasonography; respiratory distress; abdominal surgery; Age; gender; biometric; body mass index; ASA score; smoking status; history of respiratory disease
MeSH Terms: conditions — Dyspnea; Coitus; Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Abdominal laparoscopic surgery (C group) (Experimental)
  Interventions: Procedure: Diaphragmatic amplitude measurement
- Abdominal surgery by laparotomy (L group) (Experimental)
  Interventions: Procedure: Diaphragmatic amplitude measurement
- Head and neck surgery (O group) (Experimental)
  Interventions: Procedure: Diaphragmatic amplitude measurement

INTERVENTIONS:
Procedure: Diaphragmatic amplitude measurement — Diaphragmatic amplitude is measured by M Mode ultrasonography the day before and after surgery

SUMMARY:
Diaphragmatic dysfunction (DD) is one of the main risk factors for post operative respiratory distress syndrome. Ultrasonography is a diagnosis tool for DD but few studies have been published. The aim of this prospective study is to compare the achievement of diaphragmatic function depending on the type of surgery (abdominal and head and neck surgery).

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Upper abdominal or head and neck surgery
* written consent

Exclusion Criteria:

* Age <18 years
* Pregnancy
* History of neuropathy or myopathy,
* History of diaphragm paralysis, thoracic surgery, pneumothorax, pneumomediastinum

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2012-10; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Comparison of diaphragmatic amplitude measured by M-Mode ultrasonography performed the day before and the day after surgery in 3 groups: laparoscopic abdominal surgery, abdominal surgery by laparotomy and head and neck surgery. | two months

SECONDARY OUTCOMES:
All cause morbidity | within the first 28 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Département d'Anesthésie Hôpital de la Croix Rousse, Lyon, Lyon, France